CLINICAL TRIAL: NCT00109317
Title: A Phase IIIb, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Multicenter Study to Evaluate the Safety of 1.0 mg/kg Subcutaneously Administered Efalizumab in Adults With Moderate to Severe Plaque Psoriasis Who Are Candidates for Systemic Therapy
Brief Title: A Study to Evaluate Raptiva in Adults With Moderate to Severe Plaque Psoriasis Who Are Candidates for Systemic Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACD2600g
Record Dates: First submitted 2005-04-27; First posted 2005-04-27 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Psoriasis
Keywords: Moderate Plaque Psoriasis; Severe Plaque Psoriasis; Topical
MeSH Terms: conditions — Psoriasis | interventions — efalizumab

INTERVENTIONS:
Drug: Raptiva (efalizumab)

SUMMARY:
This is a Phase IIIb, randomized, double-blind, parallel-group, placebo-controlled, multicenter study designed to evaluate the safety and tolerability of efalizumab administered subcutaneously at weekly doses of 1.0 mg/kg in subjects with moderate to severe plaque psoriasis who are candidates for systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Plaque psoriasis covering >=10% of total BSA
* Diagnosis of plaque psoriasis for at least 6 months
* Minimal PASI score of 12.0 at screening
* In the opinion of the investigator, candidate for systemic therapy for psoriasis who has not been previously treated (naive to systemic treatment) or prior treatment with systemic therapy for psoriasis (e.g., PUVA, cyclosporine, corticosteroids, methotrexate, oral retinoids, MMF, thioguanine, hydroxyurea, sirolimus, azathioprine, 6-MP, etanercept)
* Body weight of <=140 kg
* 18 to 75 years old
* For women of childbearing potential, willingness to use an acceptable method of contraception to prevent pregnancy for the duration of the study
* Willingness to hold sun exposure reasonably constant and to avoid use of tanning booths or other UV light sources during the study
* Willingness to enter Study ACD2601g

Exclusion Criteria:

* Guttate, erythrodermic, or pustular psoriasis as sole or predominant form of psoriasis
* History of severe allergic or anaphylactic reactions to humanized monoclonal antibodies or fusion proteins that contain an Ig Fc region
* Clinically significant psoriasis flare during screening or on the day of randomization
* History of or ongoing uncontrolled bacterial, viral, fungal, or atypical mycobacterial infection
* History of opportunistic infections (e.g., systemic fungal infections, parasites)
* Seropositivity for human immunodeficiency virus (HIV)
* Pregnancy or lactation
* WBC count <4000/uL or >14,000/uL
* Seropositivity for hepatitis B or C virus
* Hepatic enzymes >=3x the upper limits of normal (ULN)
* History of active tuberculosis (TB) or currently undergoing treatment for TB
* Presence of malignancy within the past 5 years, including lymphoproliferative disorders
* Previous treatment with efalizumab (anti-CD11a)
* Diagnosis of hepatic cirrhosis, regardless of cause or severity
* Serum creatinine >=2x the ULN
* Hospital admission for cardiac disease, stroke, or pulmonary disease within the last year
* History of substance abuse within the last 5 years
* Any medical condition that, in the judgment of the investigator, would jeopardize the subject's safety following exposure to study drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 686 (Actual)
Dates: Start 2002-09; Study Completion 2003-02 (Actual)